CLINICAL TRIAL: NCT07264179
Title: Tracheal Cuff Pressure and Postoperative Complications: Prospective Observational Study.
Brief Title: Tracheal Cuff Pressure and Postoperative Complications: A Prospective Observational Study.
Acronym: TCP-POC
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: UNIVERSIDADE FEDERAL DO RIO GRANDE DO SUL (UFRGS) (Unknown)
Responsible Party: Principal Investigator, Andre Prato Schmidt, MD, PhD, Hospital de Clinicas de Porto Alegre
Other Study IDs: 92008125.9.0000.5327
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Tracheal Intubation; Postoperative Complications (Cardiopulmonary)
Keywords: Tracheal cuff pressure; Tracheal mucosal lesions; Cough; Orotracheal tube; Postoperative hoarseness; Pharyngolaryngeal pain; Hemoptysis
MeSH Terms: conditions — Postoperative Complications; Cough; Hemoptysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Group - Elective Surgical Patients: Single Group - Elective Surgical Patients (All patients undergoing elective surgeries with general anesthesia and orotracheal intubation; no arms as it is observational).

SUMMARY:
This prospective observational study aims to identify risk factors for tracheal mucosal injuries caused by orotracheal tube use during the intraoperative period in patients undergoing elective surgeries at the Hospital de Clínicas de Porto Alegre. The study will recruit patients sequentially for elective procedures requiring general anesthesia and orotracheal intubation. Primary outcomes include symptoms such as hoarseness, pharyngolaryngeal pain, cough, and hemoptysis, assessed up to 30 days post-surgery. A risk score for tracheal injuries will be derived.

DETAILED DESCRIPTION:
Orotracheal tubes are widely used in medical practice to secure the airway and enable invasive mechanical ventilation. Modern tubes are made of medical-grade PVC with an inflatable cuff at the distal end to isolate the lower airway, prevent gas leaks from ventilation, and reduce contamination risks from upper airway secretions or gastric content. Although current cuffs are high-volume, low-pressure, overinflation complications are common, leading to variable severity lesions (isolated or confluent lesions, tracheal mucosal edema, erosions, or ulcerations with bleeding), and symptoms like dysphonia/aphonia (15-80%), cough, pain, and hemoptysis (10-15%). Overinflation can compromise tracheal mucosal perfusion, causing ischemia, necrosis, tracheoesophageal fistulas, or tracheal rupture, especially in patients requiring prolonged intubation. Even short exposures (hours) can cause significant lesions. Many physicians rely on manual palpation or experience to set cuff pressure, often inaccurately. This study will evaluate risk factors in elective surgical patients at HCPA, using multivariate regression to identify independent variables and derive a risk score.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years.
* Patients scheduled for elective procedures requiring general anesthesia and orotracheal intubation.

Exclusion Criteria:

* Age less than 18 years.
* Refusal to participate in the study.
* Surgeries performed on an urgent or emergency basis.
* Surgeries in pregnant women.
* Cardiac surgeries.
* Surgeries requiring single-lung ventilation.
* Head and neck surgeries.
* Surgeries on the cervical segment of the dorsal spine.
* Surgeries requiring lateral or prone positioning.
* Anticipated difficult airway (unanticipated difficult airways will be included).
* Insufficient fasting time.
* Surgeries in patients admitted to intensive care units.
* Patients presenting the same symptoms included in the outcomes to be measured (pre-existing hoarseness, pain, cough, hemoptysis).
* Tracheostomized patients or those with previous tracheobronchial segment lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective procedures requiring general anesthesia and orotracheal intubation.
Sampling Method: Non-Probability Sample
Enrollment: 362 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Presence of Tracheal Injury Symptoms (Composite Outcome). | First 24 hours post-op to 30 days post-op
  Composite of hoarseness, pharyngolaryngeal pain, cough, and hemoptysis related to orotracheal tube use during surgery. Hoarseness, pain, and cough assessed via verbal numerical scale (0 = absent, 10 = worst possible). Hemoptysis assessed as present/absent, and volume (>100 ml/24h considered massive).

SECONDARY OUTCOMES:
Independent Variables for Tracheal Complications. | Intraoperative and up to 30 days post-op.
  Identification of independent variables (e.g., sex, age, tube duration, tube diameter, intubation attempts, unanticipated difficult airway, surgical table position, vasopressor use, comorbidities like hypertension, myocardial infarction, diabetes, peripheral arterial disease).

CONTACTS AND LOCATIONS:
Overall Officials: Clovis Tadeu Bevilacqua Filho, MD, MSc., Principal Investigator — Serviço de Anestesia e Medicina Perioperatória, HCPA.; Andre P Schmidt, MD, PhD, Study Chair — Serviço de Anestesia e Medicina Perioperatória, HCPA.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers in its complete form. However, an anonymized database with partially included data can be shared with others if requested and for scientific purposes (including editorial requests). The data collected will be stored in REDCap and archived securely in an appropriate location, and will not be used for any purpose other than the objectives proposed by the project. All participants in the study will sign a term of commitment for the use of institutional data.

REFERENCES:
- [Result] Grant T. Do current methods for endotracheal tube cuff inflation create pressures above the recommended range? A review of the evidence. J Perioper Pract. 2013 Dec;23(12):292-5. doi: 10.1177/175045891302301205. PMID 24404708
- [Result] Liu J, Zhang X, Gong W, Li S, Wang F, Fu S, Zhang M, Hang Y. Correlations between controlled endotracheal tube cuff pressure and postprocedural complications: a multicenter study. Anesth Analg. 2010 Nov;111(5):1133-7. doi: 10.1213/ANE.0b013e3181f2ecc7. Epub 2010 Aug 24. PMID 20736432
- [Result] Brodsky MB, Akst LM, Jedlanek E, Pandian V, Blackford B, Price C, Cole G, Mendez-Tellez PA, Hillel AT, Best SR, Levy MJ. Laryngeal Injury and Upper Airway Symptoms After Endotracheal Intubation During Surgery: A Systematic Review and Meta-analysis. Anesth Analg. 2021 Apr 1;132(4):1023-1032. doi: 10.1213/ANE.0000000000005276. PMID 33196479